CLINICAL TRIAL: NCT01852175
Title: A head-to Head Comparison of the Pharmacodynamic Effects of Prasugrel Compared With Ticagrelor in Patients With Coronary Artery Disease
Brief Title: Pharmacodynamic Effects of Prasugrel Compared With Ticagrelor in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFJ 2011-143
Record Dates: First submitted 2013-05-08; First posted 2013-05-13 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Dual antiplatelet therapy; prasugrel; ticagrelor
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel (Active Comparator): Prasugrel 60mg loading dose and 10 mg maintenance dose
  Interventions: Drug: Prasugrel
- Ticagrelor (Active Comparator): Ticagrelor 180mg loading dose and 90mg bid maintenance dose
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 60mg loading dose and 10mg maintenance dose
  Other Names: Effient
  Arms: Prasugrel
Drug: Ticagrelor — Ticagrelor 180mg loading dose and 90mg bid maintenance dose
  Other Names: Brillinta
  Arms: Ticagrelor

SUMMARY:
Recently, two P2Y12 receptor inhibitors have been approved for clinical use: prasugrel and ticagrelor. Both prasugrel and ticagrelor have shown to be associated with more potent antiplatelet effects compared with clopidogrel and are associated with an improved net clinical benefit. However, to date there are limited head-to-head comparisons of these two new agents.

DETAILED DESCRIPTION:
Dual antiplatelet therapy consisting of aspirin and clopidogrel is the cornerstone of treatment for prevention of thrombotic events in patients with coronary artery disease (CAD) undergoing percutaneous coronary intervention (PCI). However, there are a considerable number of patients who continue to have recurrent ischemic events despite this treatment regimen. These observations underscore the need for more potent antiplatelet therapies. Recently, two P2Y12 receptor inhibitors have been approved for clinical use: prasugrel and ticagrelor. Both prasugrel and ticagrelor have shown to be associated with more potent antiplatelet effects compared with clopidogrel. These more favorable pharmacodynamic effects translate into reduced ischemic event rates, at the expense of an increased risk of bleeding in patients with acute coronary syndromes. Overall, these drugs are associated with an improved net clinical benefit. These findings from large-scale clinical investigations have led to approval of prasugrel and ticagrelor. However, to date there are limited head-to-head comparisons of these two new agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known coronary artery disease
* On maintenance treatment with aspirin (81 mg per day) and clopidogrel (75 mg per day) for at least 1-month as per standard of care.
* Age between 18 and 74 years old.

Exclusion Criteria:

* History of stroke, transient ischemic attack or intracranial bleeding.
* Known allergies to aspirin, prasugrel, ticagrelor, or clopidogrel.
* Weight <60kg
* On treatment with oral anticoagulation (coumarin derivate, dabigatran).
* Hemoglobin<10 gm/dL
* Platelet count <80x106/mL
* Active bleeding or hemodynamic instability.
* Creatinine Clearance <30 mL/minute.
* Baseline ALT >2.5 times the upper limit of normal.
* Patients with sick sinus syndrome (SSS) or high degree AV block without pacemaker protection.
* Drugs interfering with 2C19 metabolism (to avoid interaction with clopidogrel): , fluconazole (Diflucan), ketoconazole (Nizoral), voriconazole (VFEND), etravirine (Intelence), felbamate (Felbatol), fluoxetine (Prozac, Serafem, Symbyax), fluvoxamine (Luvox), and ticlopidine (Ticlid).
* Drugs interfering CYP3A4 metabolism (to avoid interaction with Ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromizycin.
* Pregnant females*. *Women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Galli M, Rollini F, Been L, Zenni MM, Angiolillo DJ, Franchi F. Impact of diabetes mellitus on the pharmacodynamic effects of prasugrel and ticagrelor after switching from clopidogrel in patients with coronary artery disease. J Thromb Thrombolysis. 2022 Oct;54(3):461-469. doi: 10.1007/s11239-022-02696-4. Epub 2022 Sep 1. PMID 36048358
- [Derived] Rollini F, Franchi F, Cho JR, DeGroat C, Bhatti M, Muniz-Lozano A, Singh K, Ferrante E, Wilson RE, Dunn EC, Zenni MM, Guzman LA, Bass TA, Angiolillo DJ. A head-to-head pharmacodynamic comparison of prasugrel vs. ticagrelor after switching from clopidogrel in patients with coronary artery disease: results of a prospective randomized study. Eur Heart J. 2016 Sep 14;37(35):2722-30. doi: 10.1093/eurheartj/ehv744. Epub 2016 Feb 3. PMID 26848148

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2011 to June 2014 patients were screened at the outpatient cardiology clinics, UF Health, University of Florida, Jacksonville.
Period: Overall Study
Arm/Group | Prasugrel | Ticagrelor
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Ticagrelor | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 41 | 82
  >=65 years | 14 | 14 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 26 | 45
  Male | 36 | 29 | 65
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity by Vasodilator-stimulated Phosphoprotein (VASP)
Description: The primary end-point of the study was the comparison in the platelet reactivity index (PRI%) determined by vasodilator-stimulated phosphoprotein (VASP) at 1 week between prasugrel and ticagrelor.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: PRI%
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 55 | 55
PRI% | 32.1 (2.5) | 32.6 (2.7)

2. Secondary Outcome: Platelet Reactivity Measured by Vasodilator-stimulated Phosphoprotein (VASP)
Description: A secondary outcome was the comparison between groups of platelet reactivity index (PRI) measured by vasodilator-stimulated phosphoprotein (VASP) at 2 hours after loading dose.
Time Frame: 2 hours
Measure: Least Squares Mean (Standard Error); unit: PRI%
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 55 | 55
PRI% | 13.4 (2.7) | 15.6 (3)

3. Secondary Outcome: Platelet Reactivity Measured by Vasodilator-stimulated Phosphoprotein (VASP)
Description: A secondary outcome was the comparison between groups of platelet reactivity index (PRI) measured by vasodilator-stimulated phosphoprotein (VASP) at 24 hours after loading dose.
Time Frame: 24 hours
Measure: Least Squares Mean (Standard Error); unit: PRI%
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 55 | 55
PRI% | 14.2 (2.2) | 26.4 (2.2)

ADVERSE EVENTS:
Time Frame: 1 week
Description: Adverse events, including bleeding, bradyarrhythmias, and dyspnea, defined according to previously reported criteria were recorded
Arm/Group | Prasugrel | Ticagrelor
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 5/55
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel (N=55) | Ticagrelor (N=55)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) — Dyspnea resolved spontaneously within 24 hours

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No